CLINICAL TRIAL: NCT05746000
Title: A Nutrition Education Module to Modify Sugar Consumptions Among Individuals With Cardio Metabolic Risks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Barakatun Nisak Bt Mohd Yusof, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: My Smart Sugar Study
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Participants in the control group will attend three standard diet counselling.
  Interventions: Behavioral: Control Group (CG)
- Intervention Group (Other): Participants in the intervention group will attend three individual diet counselling and will be educated about sugar calculation (sugar exchange).
  Interventions: Behavioral: Intervention Group (IG)

INTERVENTIONS:
Behavioral: Intervention Group (IG) — Three individual diet counselling that includes sugar calculation (sugar exchange) (60 minutes per session) at baseline, week-4 and week-8.
  Arms: Intervention Group
Behavioral: Control Group (CG) — Three individual diet counselling (60 minutes per session) at baseline, week-4 and week-8.
  Arms: Control Group

SUMMARY:
The goal of this feasibility study is to assess the feasibility of a nutrition education module in modifying sugar consumption among individuals with cardiometabolic risk. The main questions it aims to answer are:

* Is the nutrition education (focusing on modifying sugars intake) intervention feasible to individuals with cardiometabolic risk?
* Can the intervention be delivered as planned and works as intended?
* What are the experiences, perspective and barriers of individuals with cardiometabolic risk when receiving the nutrition education intervention?
* Is the nutrition education intervention efficient in modifying the eating behaviour including the sugar consumption among individuals with cardiometabolic risk?

Participants in the Control Group and Intervention Group will attend three standard diet counselling, with additional sugar education for the Intervention Group.

DETAILED DESCRIPTION:
This study aims to assess the feasibility of a nutrition education module in modifying sugar consumption among individuals with cardiometabolic risk. This feasibility study will recruit patients from the Teaching Hospital of Universiti Putra Malaysia. Subjects' selection will be based on the inclusion and exclusion criteria of the study. This is a three-month feasibility study. Participants will be randomly assigned into two groups (Control and Intervention Groups). Participants in the Control Group will attend three standard diet counselling at baseline, week-4, and week-8. Participants in the Intervention Group will also attend three individual diet counselling and will be educated about sugar calculation (sugar exchange).

ELIGIBILITY:
Candidates will be screened for:

* Cardiometabolic risk factors (waist circumference, blood pressure, fasting blood glucose, triglyceride and high-density lipoprotein cholesterol)
* Pregnancy or breast feeding
* Mental health status
* Daily total sugar intake

Inclusion Criteria:

* Malaysian citizen
* patients in Teaching Hospital of Universiti Putra Malaysia
* aged 18-65 years old;
* able to read, write and communicate either in Malay or English
* education level of secondary school and above
* able to use computer or gadgets (self-reported) with internet access at home
* presence with cardiometabolic risk, defines as at least any three out of five risk factors based on:-

  1. waist circumference (men: ≥90cm, women: ≥80 cm) or;
  2. blood pressure (≥130/85 mmHg) or;
  3. having diabetes mellitus or fasting blood sugar (≥5.6mmol/L) or;
  4. triglyceride (≥1.7 mmol/L) or;
  5. high-density lipoprotein (men: <1.03 mmol/L, women: <1.3 mmol/L)
* If on medication, on stabilised dose for at least 2 months before recruitment to the study
* Daily free sugar intake ≥5% of the daily energy intake

Exclusion Criteria:

* Diagnosed with mental illness (depression, bipolar disorder, schizophrenia, dementia)
* Uncontrolled type 2 diabetes defines as HbA1c of more than 8% or hypertriglyceridemia of >10 mmol/L
* Presence of chronic diseases-related complications such as liver disease or stage 3 chronic kidney disease
* Reported abnormal thyroid-stimulating hormones
* On cancer therapy
* Having lower limb disabilities
* Breastfeeding, pregnancy, or the desire to become pregnant in the next 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible potential candidates who agree to participate in the study | At screening period. All subjects who agree to participate in the intervention will be determined.
  This can be determined by dividing the number of potential patients who agree to participate in the study by the total number of eligible patients in the patient lists.
Proportion of subjects in the intervention group who take up the intervention | At baseline of the intervention. All subjects who attend the intervention at baseline will be determined.
  This can be determined by dividing the subjects the intervention group who take up the intervention by the number of subjects who are randomly assigned to the intervention group.
Proportion of subjects who withdraw from the study or are lost to follow-up | Three months of the intervention. All subjects who withdraw from the study or are lost to follow-up throughout the three months intervention will be determined.
  This can be determined by dividing the subjects who withdraw from the study or are lost to follow-up throughout the intervention by the total number of subjects who participate in the study at baseline.

SECONDARY OUTCOMES:
Weight, height and Body Mass Index (BMI) | At baseline and week-12 of the intervention
  Weight (kilograms) and height (meters) will be combined to report BMI (kg/m2). BMI will be calculated using formula [weight in kilograms/ (height in meters)2] and cut-off point for normal BMI (18.5-24.9 kg/m2) will be used.
Waist circumference, hip circumference and waist-to-hip ratio | At baseline and week-12 of the intervention
  Waist (centimeters) and hip circumference (centimeters) will be combined to report waist-to-hip ratio. Waist-to-hip ratio will be calculated using formula (waist circumference in cm/hip circumference in cm).
Dietary intake | At baseline, week-4, week-8 and week-12 of the intervention.
  A 3-day Food Record will be used to determine the dietary intake.
Dietary sugar intake | At baseline and week-12 of the intervention.
  A semi-quantitative Food Frequency Questionnaire of added sugar intake will be used to determine the dietary sugar intake.
Eating behaviour | At baseline and week-12 of the intervention
  Eating behaviour will be determined using the Dutch Eating Behaviour Questionnaire (DEBQ), which will be evaluated based on a Likert scale with a scoring system identified as: 1 = never, 2 = seldom, 3 = sometimes, 4 = often, and 5 = very often.
Health belief | At baseline and week-12 of the intervention
  Health belief level will be determined using a Health Belief Model questionnaire, which will be evaluated based on a five Likert scale where the lowest score refers to strongly disagree, followed by disagree, neutral, agree and strongly agree.
Physical activity level | At baseline and week-12 of the intervention
  Physical activity level will be measured using International Physical Activity Questionnaire (IPAQ). And the level will be categorised as low, moderate or high.
Knowledge level | At baseline and week-12 of the intervention
  Knowledge level of healthy diet and sugar will be determined using the questions adapted from the Knowledge Assessment Questionnaire.
Blood pressure | At baseline and week-12 of the intervention
  Blood pressure will be obtained from subjects' record in the Teaching Hospital of Universiti Putra Malaysia.
Fasting blood glucose | At baseline and week-12 of the intervention
  Fasting blood glucose will be obtained from subjects' record in the Teaching Hospital of Universiti Putra Malaysia.
Triglyceride | At baseline and week-12 of the intervention
  Triglyceride level will be obtained from subjects' record in the Teaching Hospital of Universiti Putra Malaysia.
LDL-cholesterol | At baseline and week-12 of the intervention
  LDL-cholesterol level will be obtained from subjects' record in the Teaching Hospital of Universiti Putra Malaysia.
Insulin level | At baseline and week-12 of the intervention
  Insulin level will be obtained from subjects' record in the Teaching Hospital of Universiti Putra Malaysia.
Reach (participation rate) | At baseline, week-4, week-8 and week-12 of the intervention
  The participation rate will be determined by dividing the number of subjects who attend the session by the total number of subjects in the study.
Fidelity (quality of the program delivered) | At baseline, week-4, week-8 and week-12 of the intervention
  It will be measured based on observation and test account. For the diet counselling sessions, a score will be calculated to reflect the proportion of intended sessions that are delivered as scheduled. Also, a seven-item form will be used to assess whether the intended content of diet counselling is delivered. A test account will be used to monitor the message reminders received by the participants.
Dose received (what participants received) | At week-12 of the intervention
  A self-reported evaluation survey and semi-structured interview will be conducted to measure the dose received. The participants will complete an evaluation survey immediately after the intervention to assess the usefulness and satisfaction of the intervention. A semi-structured interview will be conducted to determine the usefulness of intervention components, barriers to participation, and suggestions for improvements.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No